CLINICAL TRIAL: NCT05963204
Title: A Randomized, Double-blinded, Split-face, Comparative Study to Evaluate the Synergistic Effects for Improving the Aging Midface When Pairing a Biostimulator with a Skincare Regimen
Brief Title: A Study to Evaluate the Effects for Midface Improvement When Pairing a Biostimulator with a Skincare Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.023
Record Dates: First submitted 2023-06-29; First posted 2023-07-27 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Photodamaged Skin; Volume Deficiency of the Midface
MeSH Terms: interventions — New-Fill

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Biostimulator and Facial Moisturizer A (Active Comparator): Biostimulator is sterile dry powder poly L-lactic acid with sodium carboxymethylcellulose, non-pyrogenic mannitol. Mode of administration: injection. Dosage: at investigator's discretion for optimal outcome. Frequency and duration: injection at baseline and at week 6.
  Facial Moisturizer A is a cream with active TriHex technology. Mode of administration: topical application. Frequency and duration: twice daily on half of the face for the entire study.
  Interventions: Combination Product: Sculptra and Alastin Restorative Skin Complex
- Biostimulator and Facial Moisturizer B (Active Comparator): Biostimulator is sterile dry powder poly L-lactic acid with sodium carboxymethylcellulose, non-pyrogenic mannitol. Mode of administration: injection. Dosage: at investigator's discretion for optimal outcome. Frequency and duration: injection at baseline and at week 6.
  Facial Moisturizer B is a neutral, oil-free moisturizing lotion. Mode of administration: topical application. Frequency and duration: twice daily on half of the face for the entire study.
  Interventions: Combination Product: Sculptra and CeraVe Daily Moisturizing Lotion

INTERVENTIONS:
Combination Product: Sculptra and Alastin Restorative Skin Complex — Biostimulator and cosmetics
  Arms: Biostimulator and Facial Moisturizer A
Combination Product: Sculptra and CeraVe Daily Moisturizing Lotion — Biostimulator and cosmetics
  Arms: Biostimulator and Facial Moisturizer B

SUMMARY:
To assess skin structural change in midface after treatment with a biostimulator using Line-Field Optical Coherence Tomography

DETAILED DESCRIPTION:
This is a randomized, double-blinded, split-face, comparative study.

This study is designed to enroll and randomize approximately 20 subjects. All subjects are to have midface volume loss and contour deficiency and facial photodamage.

Eligible subjects are randomized to receive study skincare products for pre-conditioning, 2 weeks before Baseline. All subjects receive biostimulator treatment at the midface by the Treating Investigator at Baseline. The method of injection is at the discretion of the Treating Investigator. A sufficient amount of product is injected to achieve optimal correction of the midface, in the opinion of the Treating Investigator.

At the 6-week visit, after all study procedures for the visit are completed, treated subjects received a second biostimulator treatment to achieve optimal aesthetic improvement. At the 12-week and 18-week visits, similar study procedures are performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with symmetrical, moderate-to-severe cheek wrinkles on each side of the face as assessed via the Galderma Cheek Wrinkles Scale.
* Subjects with symmetrical, mild-to-severe photodamage at both sides of the midface.
* Subject who in the opinion of the treating investigator would need 2 biostimulator treatments for optimal clinical outcomes.
* Ability of giving consent for participation in the study.
* Agreement to adhere to the procedures and requirements of the study and to report to the institute on the day(s) and at the time(s) scheduled for the assessments.

Exclusion Criteria:

* Subjects with asymmetrical severity or unidentical cheek wrinkle score between 2 sides of the cheek.
* Asymmetrical severity photodamage score between 2 sides of the midface.
* Subjects with a history of allergy or hypersensitivity to any ingredient of the treatment products.
* Previous tissue-augmenting therapy, contouring, or revitalization treatment in the face, except lips.
* Previous treatment/procedure in the face in the previous 6 months that, in the Investigator's opinion, would interfere with the study injections and/or study assessments or exposed the study subject to undue risk by study participation, or planning to undergo any of these procedures affecting the treatment area at any time during the study.
* Subjects with any medical condition that, in the opinion of the Investigator, would make the subject unsuitable for inclusion.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Structural change in midface post-treatment with a biostimulator compared to pre-treatment | 6 weeks and 18 weeks after Baseline
  Percent change in collagen fiber density using Line-Field Confocal Optical Coherence Tomography at defined timepoints compared to baseline. Collagen density is defined as a number of fibers and is measured on each side of the midface.

SECONDARY OUTCOMES:
Improvement in clinical grading score compared to pre-treatment | Baseline, at 6 weeks, 12 weeks, and 18 weeks after Baseline
  Percent change in skin parameters includes photodamage, roughness, radiance at defined timepoints compared to re-treatment. Each parameter is assessed by the Investigator on each side of the face using a 10-point Modified Griffiths' scale where 0 = none and 9 = severe.
Subject satisfaction using a self-assessment questionnaire | Baseline, at 6 weeks, 12 weeks, and 18 weeks after Baseline
  Survey where subjects are asked about their satisfaction with treatment outcome on each half of their face. A 5-point subject satisfaction questionnaire with the following responses: strongly agree, agree, neither agree nor disagree, disagree, strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Orit Markowitz, MD, Principal Investigator — Markowitz Medical
Locations (1):
- Markowitz Medicals, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No